CLINICAL TRIAL: NCT04391309
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Effect of Anti-CD14 Treatment in Hospitalized Patients With COVID-19
Brief Title: COVID-19 and Anti-CD14 Treatment Trial
Acronym: CaTT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped to slow rate of enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Washington (Other); Implicit Bioscience (Industry); Vanderbilt University Medical Center (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT COVID-19-003; NIAID CRMS ID#: 38756 (Other: DAIT NIAID); UM1AI109565 (NIH)
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Coronavirus Disease 2019 (COVID-19); Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Keywords: anti-CD14 (anti-CD14 chimeric monoclonal antibody); randomized double-blind placebo-controlled clinical trial; hospitalized patients
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo consists of identical-appearing diluent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- anti-CD14 + SOC (Experimental): Anti-CD14: Anticipated 150 participants randomized to 4 mg/kg on Day 1, 2 mg/kg on Days 2-4 intravenously.
  Standard of Care (SOC): All participants will receive remdesivir (antiviral) according to current approved dosing for COVID-19 illness.
  Interventions: Biological: anti-CD14; Drug: remdesivir
- Placebo + SOC (Placebo Comparator): Anticipated 150 participants randomized to Placebo diluent on Days 1-4 intravenously.
  Standard of Care (SOC): All participants will receive remdesivir (antiviral) according to current approved dosing for COVID-19 illness.
  Interventions: Other: Placebo; Drug: remdesivir

INTERVENTIONS:
Biological: anti-CD14 — 4 mg/kg on Day 1, 2 mg/kg on Days 2-4 administered intravenously (IV)
  Other Names: monoclonal antibody to CD14; IC14
  Arms: anti-CD14 + SOC
Other: Placebo — Placebo administered intravenously on Days 1-4
  Other Names: Placebo for anti-CD14
  Arms: Placebo + SOC
Drug: remdesivir — Remdesivir administered intravenously for 5 days beginning with a 200 mg loading dose on Day 1, followed by 100 mg/day on Days 2-5.
  Other Names: Veklury®

SUMMARY:
This study aims to address the following objectives:

1. To determine the efficacy of IC14, an anti-CD14 chimeric monoclonal antibody, in patients hospitalized with respiratory disease and hypoxemia due to SARS-CoV-2, in terms of improving the time to resolution of disease.
2. To determine the efficacy of IC14 in reducing the severity of respiratory disease in patients hospitalized with respiratory disease due to SARS-CoV-2.
3. To determine the safety of IC14 in patients hospitalized with respiratory disease due to SARS-CoV-2.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study of IC14, an antibody to CD14, in reducing the severity of respiratory disease in hospitalized Coronavirus Disease 2019 (COVID-19) patients.

Participants will be randomized to IC14 or matching placebo and followed for 60 days after randomization. The study drug will be administered daily on Days 1-4 by intravenous infusion. All participants will receive standard of care antiviral therapy with remdesivir.

ELIGIBILITY:
Inclusion Criteria:

Patients included in the study must meet all the following criteria:

* Patient or legally authorized representative able to provide informed consent
* Presence of SARS-CoV-2 infection documented by positive RT-PCR testing or history of positive RT-PCR test for SARS-CoV-2 within 7 days of screening
* Radiologic findings compatible with diagnosis of SARS-CoV-2 pulmonary infection
* Hypoxemia as defined by any of the following:

  * SpO2 ≤94% on room air, or
  * Requirement for ≥2L/m O2 per standard nasal cannula to maintain SpO2≥94%, but not requiring high-flow nasal cannula (defined as ≥30 L/m), and
* Negative pregnancy test for women of childbearing potential and, must be willing to use birth control for the duration of the study.

Exclusion Criteria:

An individual fulfilling any of the following criteria should be excluded from enrollment in the study:

* Receiving non-invasive positive-pressure ventilation through nasal mask, face mask, or nasal plugs
* Receiving invasive mechanical ventilation
* Patient, surrogate, or physician not committed to full support

  --Exception: a participant will not be excluded if he/she would receive all supportive care other than attempts at resuscitation from cardiac arrest)
* Anticipated survival <48 hours
* Underlying malignancy, or other condition, with estimated life expectancy of less than two months
* Significant pre-existing organ dysfunction prior to randomization

  * Lung: Currently receiving home oxygen therapy as documented in medical record
  * Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record
  * Renal: End-stage renal disease requiring renal replacement therapy or eGFR <30 mL/min
  * Liver: Severe chronic liver disease defined as Child-Pugh Class C or AST or ALT >5x upper limit of normal
  * Hematologic: Baseline platelet count <50,000/mm^3
* Presence of co-existing infection, including, but not limited to:

  * HIV infection not virally suppressed and with pre-hospitalization CD4 counts ≤ 500 cell/mm^3
  * Active tuberculosis or a history of inadequately treated tuberculosis
  * Active hepatitis B or hepatitis C viral infection
* Ongoing immunosuppression

  * Solid organ transplant recipient
  * High-dose corticosteroids (equivalent to >20 mg/prednisone/day) within the past 28 days, except for dexamethasone except for dexamethasone or equivalent treatment for COVID-19 illness
  * Oncolytic drug therapy within the past 14 days
* Current treatment, or treatment within 30 days or five half-lives (whichever is longer) with etanercept (Enbrel®), infliximab (Remicade®), adalimumab (Humira®), certolizumab (Cimzia®), golimumab (Simponi®), anakinra (Kineret®), rilonacept (Arcalyst®), tocilizumab (Actemra®), sarilumab (Kevzara®), siltuximab (Sylvant®), or other potent immunosuppressant or immunomodulatory drugs or treatments
* Current treatment with an anti-viral medication for COVID-19 (e.g. hydroxychloroquine, lopinavir/ritonavir), other than remdesivir
* Current enrollment in an interventional trial for COVID-19
* History of hypersensitivity or idiosyncratic reaction to IC14
* Women who are currently breastfeeding
* Received a live-attenuated vaccine within 30 days prior to enrollment
* Received five or more doses of remdesivir, including the loading dose, outside of the study as treatment for COVID-19, or
* Any condition that in the opinion of the treating physician will increase the risk for the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Wurfel, MD, PhD, Study Chair — University of Washington: Division of Pulmonary, Critical Care and Sleep Medicine; Thomas R. Martin, MD, Study Chair — University of Washington: Division of Pulmonary, Critical Care and Sleep Medicine
Locations (5):
- United States (5):
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center-Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institutes of Health News Release Describing Study — https://www.nih.gov/news-events/news-releases/nih-trial-anti-cd14-antibody-treat-covid-19-respiratory-disease-begins
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: NIAID Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Centers for Disease Control and Prevention -COVID-19 resources — https://www.cdc.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 participants were enrolled across 5 US sites from April 2021 to January 2022. Of these enrolled, 41 participants were randomized and 40 initiated study treatment. 8 enrolled participants were not randomized because they did not meet eligibility criteria, and one randomized participant did not initiate study treatment because they withdrew their consent.
Pre-assignment Details: 8 enrolled participants were not randomized because they did not meet eligibility criteria.
Groups:
- IC14: Subjects received IC14 4 mg/kg intravenously on Day 1, followed by IC14 2 mg/kg/day intravenously on Days 2-4 (totaling 4 consecutive days). Subjects also received remdesivir 200 mg intravenously on Day 1, followed by 100 mg intravenously daily on Days 2-5 (totaling 5 consecutive days).
- Placebo: Subjects received 0.9% w/v Sodium Chloride in a matching bag and volume administered intravenously daily on Days 1-4 (totaling 4 consecutive days). Subjects also received remdesivir 200 mg intravenously on Day 1, followed by 100 mg intravenously daily on Days 2-5 (totaling 5 consecutive days).
Period: Overall Study
Arm/Group | IC14 | Placebo
Started | 21 | 20
Included in the Modified Intent to Treat Population (miTT) | 20 | 20
Completed | 15 | 15
Not Completed | 6 | 5
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat population (mITT), that included all participants who were randomized and treated with at least one dose of investigational product. Measures reflect the assessment of clinical status at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | IC14 | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (14.7) | 47.1 (13.6) | 50.85 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 13 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 15 | 15 | 30
  Other | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Assessment of Clinical Status According to Eight-Point Ordinal Scale [Count of Participants; unit: Participants] — The Eight-Point Ordinal Scale - assessment of the clinical status at baseline:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen; no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen; requiring ongoing medical care
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or ECMO
  8. Death
  Participants
    1 | 0 | 0 | 0
    2 | 0 | 0 | 0
    3 | 0 | 0 | 0
    4 | 1 | 4 | 5
    5 | 18 | 14 | 32
    6 | 1 | 2 | 3
    7 | 0 | 0 | 0
    8 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Time to Clinical Recovery, Defined as the Time From Baseline to the First Day That Subject is in Categories 1, 2, or 3 on the Eight-Point Ordinal Scale Through Day 28.
Description: The Primary Endpoint is time to clinical recovery, defined as the time from baseline to the first day that a subject is in categories 1, 2, or 3 on the Eight-Point Ordinal Scale through Day 28 (range 1 [best] to 8 [worst]). The Eight-Point Ordinal Scale is an assessment of the clinical status on each study day. The Scale is defined as follows:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Hospitalized, not requiring supplemental oxygen-no longer requires ongoing medical care
  4. Hospitalized, not requiring supplemental oxygen-requiring ongoing medical care (COVID-19-related or otherwise)
  5. Hospitalized, requiring supplemental oxygen
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  8. Death
Time Frame: Within the 28 day period following baseline
Population: Modified Intent to Treat population (mITT), that included all participants who were randomized and treated with at least one dose of investigational product.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
days | 6 [5 to 11] | 5 [4 to 10]
Statistical Analysis 1: Comparison: IC14 vs Placebo; Test type: Superiority; p = 0.435, Log Rank

2. Secondary Outcome: Days Alive and Free of Any Episodes of Acute Respiratory Failure Through Day 28
Description: Episodes of acute respiratory failure are defined as by need for the following oxygen delivery resources:
  1. High-flow nasal cannula (flow rates ≥30L/min with FiO2 ≥0.4)
  2. Noninvasive positive-pressure ventilation through nasal or face mask, or nasal plugs
  3. Endotracheal intubation and mechanical
  4. Extracorporeal membrane oxygenation
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  0 days | 1 | 1
  24 days | 1 | 0
  27 days | 0 | 1
  28 days | 18 | 18
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact

3. Secondary Outcome: Change in the Ordinal Scale From Baseline to Day 14
Description: A larger negative change indicates a greater improvement in clinical status from baseline. The Eight-Point Ordinal Scale is an assessment of the clinical status on each study day (1 is best, 8 is worst). The Scale is defined as follows:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen.
  3. Hospitalized, not requiring supplemental oxygen; no longer requires ongoing medical care.
  4. Hospitalized, not requiring supplemental oxygen; requiring ongoing medical care (COVID-19-related or otherwise).
  5. Hospitalized, requiring supplemental oxygen.
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices.
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  8. Death.
Time Frame: Within the 14 day period following baseline.
Population: Modified Intent to Treat population (mITT), that included all participants who were randomized and treated with at least one dose of investigational product, who additionally had data collected on Day 14.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -3.1 (1.6) | -2.8 (1.6)
Statistical Analysis 1: Comparison: IC14 vs Placebo; Test type: Superiority; p = 0.391, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Ordinal Scale From Baseline to Day 28.
Description: as for outcome 3
Time Frame: Within the 28 day period following baseline.
Population: Modified Intent to Treat population (mITT), that included all participants who were randomized and treated with at least one dose of investigational product, who additionally had data collected on Day 28.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 15 | 16
units on a scale | -3.7 (0.6) | -3.3 (1.6)
Statistical Analysis 1: Comparison: IC14 vs Placebo; Test type: Superiority; p = 0.895, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Ordinal Scale Value on Day 14.
Description: The Eight-Point Ordinal Scale is an assessment of the clinical status on each study day (1 is best, 8 is worst). The Scale is defined as follows:
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities and/or requiring home oxygen.
  3. Hospitalized, not requiring supplemental oxygen; no longer requires ongoing medical care.
  4. Hospitalized, not requiring supplemental oxygen; requiring ongoing medical care (COVID-19-related or otherwise).
  5. Hospitalized, requiring supplemental oxygen.
  6. Hospitalized, on non-invasive ventilation or high-flow oxygen devices.
  7. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  8. Death.
Time Frame: Day 14 following baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | 1.9 (1.6) | 2.0 (1.6)
Statistical Analysis 1: Comparison: IC14 vs Placebo; Test type: Superiority; p = 0.702, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: All-Cause Mortality Through Day 28.
Description: Mortality due to all causes during the observation period.
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Alive | 19 | 20
  Died | 1 | 0
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — P-value based on Fishers exact test, which enumerates all possible tables that have same margins as observed & calculates proportion of tables where values are more extreme than observed. P-value of 1 = the observed table is the most extreme

7. Secondary Outcome: All-Cause Mortality Through Day 60.
Description: Mortality due to all causes during the observation period.
Time Frame: Within the 60 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Alive | 19 | 19
  Died | 1 | 1
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Participants Alive and Free of Any Episode of Acute Respiratory Failure Through Day 28
Description: Episodes of acute respiratory failure are defined as by need for the following oxygen delivery resources:
  1. High-flow nasal cannula (flow rates ≥30L/min with FiO2 ≥0.4)
  2. Noninvasive positive-pressure ventilation through nasal or face mask, or nasal plugs
  3. Endotracheal intubation and mechanical ventilation
  4. Extracorporeal membrane oxygenation
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Yes | 18 | 18
  No | 2 | 2
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the anlysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

9. Secondary Outcome: Days Alive and Free of Invasive Mechanical Ventilation Through Day 28
Description: Endotracheal intubation and mechanical ventilation.
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  0 days | 1 | 1
  28 days | 19 | 19
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

10. Secondary Outcome: Percentage of Participants Alive and Free of Invasive Mechanical Ventilation Through Day 28
Description: Endotracheal intubation and mechanical ventilation.
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Yes | 19 | 19
  No | 1 | 1
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

11. Secondary Outcome: Percentage of Participants Alive and Discharged From the Hospital Through Day 28
Description: Participants must be alive and discharged from hospital.
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Yes | 19 | 19
  No | 1 | 1
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

12. Secondary Outcome: Percent of Participants Who Begin Corticosteroid Therapy for Worsening COVID-19 Illness After Randomization
Description: Initiation of corticosteroid therapy.
Time Frame: Within the 28 day period following baseline.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Yes | 1 | 1
  No | 19 | 19
Statistical Analysis 1: Comparison: IC14 vs Placebo; All categories included in the analysis; Test type: Superiority; p = 1, Fisher Exact — [p-value comment as in outcome 6, analysis 1]

13. Secondary Outcome: Serious Adverse Events (SAEs)
Description: Number of serious adverse events
Time Frame: Within the 28 day period following baseline.
Population: All participants who initiated study treatment.
Measure: Number; unit: Serious Adverse Events
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Serious Adverse Events | 6 | 4

14. Secondary Outcome: Adverse Events (AEs)
Description: Number of Grade 3 and 4 clinical and/or laboratory adverse events
Time Frame: Within the 28 day period following baseline.
Population: All participants who initiated study treatment.
Measure: Number; unit: Adverse Events
Arm/Group | IC14 | Placebo
Number analyzed (Participants) | 20 | 20
Adverse Events
  Severe (Grade 3) | 12 | 10
  Life Threatening (Grade 4) | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 0 - Day 60
Description: Adverse Events were collected through Day 60
Arm/Group | IC14 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 1/20
Other Adverse Events (participants affected / at risk) | 16/20 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC14 (N=20) | Placebo (N=20)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC14 (N=20) | Placebo (N=20)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 2 (2) | 0 (0)
Dry macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 2 (2)
Incipient senile cataract (Eye disorders) | 1 (1) | 0 (0)
Lattice degeneration of retina (Eye disorders) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal macroaneurysm (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Senile nuclear sclerosis (Eye disorders) | 5 (6) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Perianal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrush (Gastrointestinal disorders) | 0 (0) | 1 (2)
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Cardiac troponin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in thigh (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Choroidal nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache tension (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Calcified lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Localized maculopapular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
The trial was terminated early because of slow recruitment and cannot be considered fully powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04391309/Prot_SAP_001.pdf